CLINICAL TRIAL: NCT04135235
Title: The Effect and Safety of Propofol Fumarate for Mother-to-child Blocking of Hepatitis B
Brief Title: Effect and Safety of Propofol Fumarate for Mother-to-child Blocking of Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wei Yi, Director, Head of Obstetrics and Gynecology, Beijing Ditan Hospital
Other Study IDs: KY2019-08
Record Dates: First submitted 2019-10-12; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis B Infection; High Viral Load
Keywords: Chronic Hepatitis B; Pregnant woman; High viral load; Tenofovir fumarate
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAF group: take propofol fumarate for Maternal and child blockade treatment
  Interventions: Drug: TAF
- TDF group: take difenofurate fumarate for Maternal and child blockade treatment
  Interventions: Drug: TDF

INTERVENTIONS:
Drug: TAF — Propofol tenofovir fumarate
  Groups: TAF group
Drug: TDF — Dipirofurate fumarate tenofovir
  Groups: TDF group

SUMMARY:
This study is a prospective study. The subject will select 440 cases of pregnant women with high hepatitis B virus load, and one group will take maternal and child blockade treatment with propofol fumarate. One group will take tenofovir disoproxil fumarate. Broken treatment, compare the failure rate of maternal and child blockade and the incidence of maternal and child adverse events in the two groups, and explore the efficacy and safety of propofol flavuril for the treatment of hepatitis B mother-infant block.

DETAILED DESCRIPTION:
This study was a prospective cohort study. Because propofolofofovir is not covered by medical insurance and is more expensive, and there are factors such as renal function damage and the risk factors that can not use tenofovir, it is difficult to conduct randomized controlled cases. The subject will select 440 cases of pregnant women with high hepatitis B virus load. After signing the informed consent form, according to the patient's wishes, one group will take the mother-infant blockade of propofol fumarate, and one group will take fumaric acid. In the case of maternal and child blockade of benifovir, the incidence of maternal and child block failure and the incidence of maternal and child adverse events were compared between the two groups, and propofol fumarate was used for maternal and child blockade of hepatitis B. The effectiveness and safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* No nucleoside analog antiviral drugs have been used in the past.
* HBsAg and HBeAg double positive, HBV DNA>106 IU/mL.
* Fully inform the risk to voluntarily join the study and sign the informed consent form.

Exclusion Criteria:

* Combine other viral infections: such as HCV, HIV, CMV, etc.;
* amniocentesis during pregnancy;
* Liver cirrhosis and liver cancer;
* Other autoimmune diseases and liver diseases;
* fetal ultrasound screening in early and middle pregnancy found deformity.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: High HBV viral load (HBV DNA ≥ 106 IU / mL) pregnant women with chronic HBV infection. All pregnant women with chronic HBV infection were in compliance with the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015).
Sampling Method: Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
the blocking successful rate of HBV mother-to-child transmission | 7 months after birth
  HBV mother-to-child transmission blocking success rate (negative HBsAg and HBV DNA negative 7 months after birth)

SECONDARY OUTCOMES:
The incidence of abnormal growth | at birth, at the 7 months after birth
  The incidence of abnormal growth at birth
The incidence of abnormal development | at birth, at the 7 months after birth
  The incidence of abnormal development at birth

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yi, Doctor, Principal Investigator — Beijing Ditan Hospital; Yao Xie, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China